CLINICAL TRIAL: NCT07152509
Title: The Effect of Body Weight on Physical Activity Level, Functional Capacity, Balance, and Quality of Life in Individuals With Type 2 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BezmialemUNV2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Body Mass Index; Functional Capacity; Balance
Keywords: quality of life; type 2 diabetes mellitus; body mass index; physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus Group: Participants diagnosed with type 2 diabetes mellitus will be included. Participants will undergo comprehensive assessment including body composition, muscle strength, hand grip strength, physical activity level, functional capacity, balance, and quality of life. No interventional procedure will be applied; the study is observational and cross-sectional.
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — The demographic, clinical, and personal characteristics of the individuals will be collected and recorded through a questionnaire. For all participants, body fat percentage (%), skeletal muscle mass percentage (%), visceral fat percentage (%), and resting metabolic rate (kcal), measured using the Omron Body Composition Monitor, will be recorded. Waist and hip circumference will be measured with a tape measure; lower extremity muscle strength (M. Quadriceps) will be assessed with a muscle hand-held dynamometer; grip strength will be assessed with a hand grip dynamometer; physical activity level will be evaluated using the International Physical Activity Questionnaire-Short Form (IPAQ-SF); functional capacity will be measured with the 6-Minute Walk Test (6MWT); postural stability and balance will be assessed with the Biodex Balance System; clinical balance will be assessed with the Berg Balance Scale; quality of life will be evaluated using the Nottingham Health Profile (NHP)

SUMMARY:
This study aims to investigate the effects of body weight on physical activity level, functional capacity, balance, and quality of life in patients with type 2 diabetes mellitus (T2DM). A total of 50 volunteer patients who meet the inclusion criteria will be recruited from the Internal Medicine and Nutrition outpatient clinics of Bezmialem Vakıf University Hospital.

Participants will be prospectively evaluated through face-to-face interviews. Assessments will include body composition analysis (Omron Body Composition Monitor), waist-to-hip ratio, lower extremity muscle strength (Muscle Hand-Held Dynamometer), grip strength (Hand Grip Dynamometer), physical activity level (International Physical Activity Questionnaire-Short Form), functional capacity (6-Minute Walk Test), balance (Biodex Balance System), clinical balance (Berg Balance Scale), and quality of life (Nottingham Health Profile).

All statistical analyses will be performed using IBM SPSS Statistics 20. With this study, we aim to comprehensively evaluate multiple parameters in individuals with T2DM and investigate their interrelationships, thereby contributing to the current body of knowledge in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Type 2 Diabetes Mellitus for at least 1 year
* Being between 18 and 65 years of age
* Having an HbA1c value between 6.5% and 11% at the time of diagnosis
* No cognitive or mental problems
* Ability to walk independently
* Willingness to participate in the study

Exclusion Criteria:

* Presence of uncontrolled cardiovascular and pulmonary disease
* Presence of vertigo or various vestibular system disorders
* Presence of severe neurological or respiratory disease
* History of stroke or myocardial infarction
* Presence of a major musculoskeletal problem
* Presence of chronic renal failure
* Presence of diabetic ulcer or neuropathy
* Pregnancy
* Presence of hemolytic or renal anemia
* Presence of serious visual, hearing, or speech impairments leading to lack of cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years with a diagnosis of Type 2 Diabetes Mellitus for at least 1 year, attending the Internal Medicine and Diet outpatient clinics, who meet the inclusion criteria and voluntarily agree to participate
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | At baseline (single assessment)
  Functional capacity will be evaluated using the 6-minute walk test (6MWT). At the beginning and end of the test, participants' oxygen saturation, heart rate, blood pressure, Borg dyspnea, and fatigue scores will be recorded. The test will be conducted in a 30-meter straight corridor, marked at 10-meter intervals, with chairs placed at both the starting and finishing points. Participants will be instructed to walk for 6 minutes at the fastest pace they can manage without running. To estimate the expected 6MWT distance, the reference equation by Enright et al. will be used in this study.
Assessment of Quality of Life Using the Nottingham Health Profile | At baseline (single assessment)
  To evaluate patients' quality of life, the Nottingham Health Profile (NHP) will be used. The scale consists of six subdomains: pain, emotional reactions, sleep, social isolation, physical mobility, and energy. Within each subdomain, a score of 0 indicates the best quality of life, while a score of 100 indicates the worst quality of life.

SECONDARY OUTCOMES:
Body Composition | At baseline (single assessment)
  For body composition analysis, the body mass index (BMI) of the participants (Body weight/height²) will be calculated. Using the Omron BF511 Body Composition Monitor (Omron Healthcare Co. Ltd; Japan), body fat percentage (%), skeletal m
waist-to-hip ratio | At baseline (single assessment)
  Waist circumference will be measured in the standing position at the level of the umbilicus during the expiratory phase using a tape measure, and recorded in centimeters ("cm"). Hip circumference will be measured in the same position at the level of the greater trochanter and recorded in centimeters ("cm"). The waist-to-hip ratio will then be calculated.
Lower Extremity Muscle Strength Assessment | At baseline (single assessment)
  Measurement of lower extremity muscle strength will be performed in a seated position, with the dominant leg in full knee extension, by applying maximum resistance using a handheld electronic dynamometer placed just above the ankle joint. The assessment will be conducted on the quadriceps muscle group using a handheld electronic dynamometer (Commander Muscle Tester; JTECH Medical, USA) and recorded in Newtons (N).
Handgrip Strength | At baseline (single assessment)
  Handgrip strength will be measured on the dominant side using a Jamar hand dynamometer and recorded in pounds (lb). The test will be performed while the patients are seated comfortably on a chair, with the shoulder in adduction and neutral position, the elbow at 90° flexion, and the forearm and wrist in a neutral position.
Physical Activity Assessment | At baseline (single assessment)
  Participants' physical activity levels will be evaluated using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). The IPAQ short form consists of seven questions designed to determine, on a daily basis over the past seven days, the time spent in vigorous physical activity (VPA), moderate physical activity (MPA), walking (W), and sitting (sedentary time). To calculate the total physical activity score, the weekly duration (minutes) of each activity is multiplied by the Metabolic Equivalent of Task (MET) values established for the IPAQ, and the resulting scores are obtained. The Turkish validity and reliability study of the IPAQ-Short Form was conducted by Sağlam M. et al.
Assessment of Functional Balance | At baseline (single assessment)
  Patients' functional balance levels will be evaluated using the Turkish version of the Berg Balance Scale (BBS). This scale consists of tasks commonly used in daily life, such as static sitting, standing balance, transfers, turning, and picking up an object from the floor. Each item is scored on a scale from 0 (unable to perform the task) to 4 (normal performance).
Postural stability assessment | At baseline (single assessment)
  Postural stability assessment will be performed using the Biodex Balance System (BBS) (Biodex Medical System, Inc; USA), including the Postural Stability Test for static postural stability and the Limits of Stability Test. The postural stability test evaluates the patient's ability to maintain their center of balance, and deviations from the center are recorded. The limits of stability test assesses the ability to move and control the center of gravity within the base of support. A higher score indicates a higher level of control.

CONTACTS AND LOCATIONS:
Overall Officials: SEMİRAMİS ÖZYILMAZ, Assoc. Prof., Principal Investigator — Bezmialem Vakıf University,Facult Of Health Sciences, Department Of Physiotherapy And Rehabilitation
Locations (1):
- Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The plan for IPD sharing has not yet been determined

REFERENCES:
- [Result] Rejeski WJ, Lang W, Neiberg RH, Van Dorsten B, Foster GD, Maciejewski ML, Rubin R, Williamson DF; Look AHEAD Research Group. Correlates of health-related quality of life in overweight and obese adults with type 2 diabetes. Obesity (Silver Spring). 2006 May;14(5):870-83. doi: 10.1038/oby.2006.101. PMID 16855197
- [Result] Awotidebe TO, Adedoyin RA, Yusuf AO, Mbada CE, Opiyo R, Maseko FC. Comparative functional exercise capacity of patients with type 2-diabetes and healthy controls: a case control study. Pan Afr Med J. 2014 Nov 7;19:257. doi: 10.11604/pamj.2014.19.257.4798. eCollection 2014. PMID 25852800